CLINICAL TRIAL: NCT01400178
Title: Cochlear Implants in Post-lingually Children: Results After 10 Years
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Liege Franzini Tanamati, Doctor, University of Sao Paulo
Other Study IDs: 186/2008
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Deafness; Hearing Impairment
Keywords: cochlear implant; children; follow up; results
MeSH Terms: conditions — Deafness; Hearing Loss

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Objectives: To assess a group of post-lingually children after 10 years of implantation with regard to speech perception, speech intelligibility, and academic/occupational status.

Study Design: A prospective transversal study. Setting: Pediatric referral center for cochlear implantation. Patients: Ten post-lingually deafened children with Nucleus and Med-El cochlear implants.

Interventions: Speech perception and speech intelligibility tests and interview.

Main Outcome Measures: The main outcome measures were score of Hint sentences recognition (silence and noise), speech intelligibility scores(write-down intelligibility and rating scale scores) and academic/ occupational status.

ELIGIBILITY:
Inclusion Criteria:

* postlingually deaf
* age at cochlear implant: < 18 years
* more than 10 years of cochlear implant use

Exclusion Criteria:

* other disabilities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The age at evaluation was 19,3 to 29,2 years. The age at cochlear implant surgery was 5,4 to 16,10 years. The etiology of the deafness was: meningitis (5), ototoxic (1), mumps (2) and unknown (2).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bionic Ear Center, São Paulo, São Paulo, Brazil